CLINICAL TRIAL: NCT02103777
Title: High Versus Low Dose of Caffeine for Apnea of Prematurity: A Double Blind Randomized Control Trial
Brief Title: High Versus Low Dose of Caffeine for Apnea of Prematurity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Associate Professor, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICU MUCH 2013
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Apnea; Preterm Infants
Keywords: high dose of caffeine; low dose of caffeine; prevention
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose caffeine (Active Comparator): High dose (loading 40 mg/kg/day equivalent to 20 mg /kg/day of caffeine base and maintenance of 20 mg/kg/day equivalent to 10 mg /kg/day of caffeine base)
  Interventions: Drug: Caffeine citrate
- Low dose caffeine (Active Comparator): Low dose (loading 20 mg/kg/day equivalent to 10 mg /kg/day of caffeine base and maintenance of 10 mg/kg/day equivalent to 5 mg /kg/day of caffeine base) caffeine.
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — Caffeine will be given by either high dose in Arm 1 or low dose in Arm 2

SUMMARY:
The optimum caffeine dose for apnea of prematurity has not been well investigated so the objective of the study is to compare high versus low dose of caffeine citrate to facilitate successful extubation in mechanically ventilated preterm infants.

DETAILED DESCRIPTION:
A randomized, double blind, clinical trial which will be conducted in Neonatal Intensive Care Unit, Mansoura University Children Hospital, Egypt on preterm infants born less than 32 weeks gestation mechanically ventilated within the first 10 days of life to study the optimum caffeine dose for apnea of prematurity and compare High dose (loading 40 mg/kg/day equivalent to 20 mg /kg/day of caffeine base and maintenance of 20 mg/kg/day equivalent to 10 mg /kg/day of caffeine base) versus low dose (loading 20 mg/kg/day equivalent to 10 mg /kg/day of caffeine base and maintenance of 10 mg/kg/day equivalent to 5 mg /kg/day of caffeine base) caffeine citrate started within the first 10 days of life and its effect on need of re-intubation within 72 hours of extubation from mechanical ventilation as primary outcome and frequency and duration of apnea, duration of mechanical ventilation and oxygen support, length of hospital stay, neonatal mortality, chronic lung disease, necrotising enterocolitis, intraventricular haemorrhage, periventricular leukomalacia, hydrocephalus, retinopathy of prematurity, and caffeine side effects as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* newborn infant less than 32 weeks gestation with the diagnosis of apnea

Exclusion Criteria:

* newborn infants with gestational age more than 32 weeks.
* newborn infant with congenital malformations or chromosomal anomalies.

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Successful extubation from mechanical ventilation | 72 hours after extubation from mechanical ventilation
  Need of re-intubation within 72 hours of extubation from mechanical ventilation

SECONDARY OUTCOMES:
Apnea of prematurity | Expected average of 8 weeks post natal age
  Frequency and documented days of apnea
Duration of mechanical ventilation and oxygen support | Expected 4 to 6 weeks postnatal age
length of hospital stay | Expected 8 weeks
Neonatal mortality | Expected 8 weeks
  Death before hospital discharge
Chronic lung disease | By 36 weeks corrected gestational age
  Need for oxygen by 36 weeks corrected gestational age
Necrotising enterocolitis | Expected 6 weeks
Intraventricular haemorrhage | Expected 2 weeks
Periventricular leukomalacia | Expected 8 weeks
Hydrocephalus | Expected 8 weeks
Retinopathy of prematurity | Expected 8 weeks
Caffeine side effects. | Expected 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: sameh m abbas, master, Principal Investigator — Mansoura University Children Hospital; nehad a nasef, MD, Study Director — Mansoura University Children Hospital
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt